CLINICAL TRIAL: NCT04151706
Title: CD34 Selected Allogeneic Hematopoietic Cell Transplantation With Myeloablative Conditioning and CD8+ Memory T Cell Infusion For Patients With Myelodysplastic Syndrome, Acute Leukemia, and Chronic Myelogenous Leukemia
Brief Title: CD34 Selected Allogeneic HCT w/ Myeloablative Conditioning Plus CD8+ Memory TCell Infusion in MDS, AL and CML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Lowsky (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Robert Lowsky, Professor of Medicine (Blood and Marrow Transplantation and Cellular Therapy), Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-49023; BMT339 (Other: OnCore); IRB-49023 (Other: Stanford IRB); P01CA049605 (NIH)
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndromes; Acute Leukemia; Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Thiotepa; fludarabine; fludarabine phosphate; Busulfan; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- fTBI/Thiotepa/fludarabine (Experimental): Participants will be infused on Day 0 with donor derived CD34+ selected cells combined with CD8+CD45RA- T cells {CD Memory T Cells} following a standard myeloablative conditioning regimen that might consist of fTBI, Thiotepa, and Fludarabine or Busulfan and Cyclophosamide.
  Interventions: Drug: CD8+ Memory T Cell Infusion; Drug: Thiotepa; Drug: Fludarabine; Radiation: Hyperfractionated TBI; Drug: Busulfan; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: CD8+ Memory T Cell Infusion — Allogeneic phenotypic CD8+ memory T cells from HLA matched donors infused at the time of hematopoietic cell transplantation
  Other Names: Enriched for CD8+CD45RA memory T cells.
Drug: Thiotepa — 5 mg/kg/day: IV for 2 consecutive days (days -6 to -5)
  Other Names: Tepadina; thiophosphamide; TESPA
Drug: Fludarabine — 25 mg/m2/day: IV for 5 consecutive days (days -6 to -2)
  Other Names: Beneflur
Radiation: Hyperfractionated TBI — Administered in 11 fractions of 125 cGy over 4 days (Total dose of 1375 cGy)
Drug: Busulfan — 6 mg/kg/dose Q24h IV. Infused over 3 hours. 1 dose per day x 4 consecutive days x 3.6 mg/kg/dose = 14.4 mg/kg
  Other Names: Busulfanum
Drug: Cyclophosphamide — 60 mg/kg/dose Q24h IV. Infused over 2 hours. 1 dose per day x 2 consecutive days x 60 mg/kg/dose = 120 mg/kg
  Other Names: Cytoxan; Neosar

SUMMARY:
This study will evaluate combining stem cells from the patient's matched sibling donor (a standard CD34-selected transplant) with a second infusion of white blood cells called "CD8 memory T-cells" from their sibling donor.

DETAILED DESCRIPTION:
Primary Objective: To determine the rate of graft versus host disease (GvHD) free, relapse free survival (GRFS) at one year following CD34 selected allogeneic hematopoietic cell transplantation using myeloablative conditioning combined with an infusion of phenotypic CD8+ memory T cells from human leukocyte antigen (HLA) matched donors for patients with myelodysplastic syndrome (MDS), acute myeloid leukemia (AML), or acute lymphoblastic leukemia (ALL) and chronic myeloid leukemia (CML).

Secondary Objective: To determine the rate of graft rejection, acute and chronic GvHD, non relapse mortality, relapse, overall survival, and disease free survival.

ELIGIBILITY:
Recipient Inclusion Criteria:

* Acute leukemia, in morphologic complete remission, OR myelodysplasia with < 10% blasts in the marrow, and no circulating blasts that contain auer rods. Patients with chronic myelomonocytic leukemia (CMML) must have a WBC count ≤ 10,000 cells/μL and < 10% blasts in the marrow.
* Planned myeloablative conditioning regimen at Stanford University Medical Center.
* Karnofsky or Lansky Performance Score ≥ 70%.
* Must have an HLA related donor as follows: onor must be an 8/8 match for HLA A, B and C at intermediate (or higher) resolution, and DRB1 at high resolution using DNA based typing. The donors must be willing to receive G CSF followed by collection of cells by apheresis, and must meet the Program's criteria for donation.
* Cardiac function: Ejection fraction at rest ≥ 40%.
* Serum creatinine value of < 1.5 mg/dL, or an estimated creatinine clearance greater than 50 mL/minute (using the Stanford calculator for eGFR available in EPIC)
* Diffusing capacity of the lungs for carbon monoxide (DLCO) ≥ 50% (adjusted for Hgb)
* Forced vital capacity (FVC) ≥ 50%.
* Forced expiratory volume (FEV1) ≥ 50%.
* Total bilirubin < 2 times the upper limit of normal (ULN) (unless the elevated bilirubin is attributed to Gilbert's Syndrome)
* Alanine aminotransferase (ALT) < 2.5 x ULN
* Aspartate aminotransferase (AST) < 2.5 x ULN
* Total bilirubin < 2 times the upper limit of normal (unless elevated bilirubin is attributed to Gilbert's Syndrome)
* Signed informed consent

Recipient Exclusion Criteria:

* Prior autologous or allogeneic hematopoietic stem cell transplant
* Prior malignancies, except resected non melanoma or treated cervical carcinoma in situ. Cancer treated with curative intent ≥ 5 years previously is allowed. Cancer treated with curative intent < 5 years previously will not be allowed unless approved by the Protocol Officer or one of the Protocol Chairs
* Active central nervous system (CNS) involvement by malignant cells
* Presence of fluid collection (ascites, pleural or pericardial effusion) that interferes with methotrexate clearance or makes methotrexate use contraindicated
* Requirement for supplemental oxygen
* Uncontrolled bacterial, viral or fungal infections (currently taking medication and with progression or no clinical improvement) at time of enrollment
* History of uncontrolled autoimmune disease or on active treatment (defined as > 5 mg prednisone daily)
* Seropositive for HIV 1 or 2
* Seropositive for HTLV I or -II
* Active Hepatitis B or C viral replication by polymerase chain reaction (PCR)
* Documented allergy to iron dextran or murine proteins
* Pregnant (positive serum or urine βHCG) or breastfeeding)
* Females of childbearing potential (FCBP) or men who have sexual contact with FCBP unwilling to use an effective form of birth control or abstinence for one year after transplantation
* Unable to comply with the treatment protocol, including appropriate supportive care, follow up and research tests.
* Planned to receive post transplant maintenance therapy except for fms-like tyrosine kinase 3 (FLT3) inhibitors or BCR ABL tyrosine kinase inhibitors (TKIs).

Donor Inclusion Criteria:

* HLA matched donor (matching at 8/8 antigens or alleles including HLA A, B, C, and -DRB1).
* ≥ 18 years to < 66.0 years
* State of general good health
* Completed a donor evaluation with history, medical examination and standard blood tests within 60 days of starting the hematopoietic cell collection procedure. In order to fairly represent the interests of the donor, the donor evaluation and consent will be performed by a study team member other than the recipient's attending physician.
* Hepatitis A, B and C, HIV 1 and 2, HTLV, VZV, EBV, HSV, West Nile virus, Syphilis Treponema, T cruzi (Chagas), CMV, and the MPX NAT IDT (HIV/HCV/HBV) will be tested as per national standard of care guidelines for transplant donors. Donors who are HIV positive will be excluded. Donors who are positive by serology for Hepatitis B or C are eligible as long as PCR for RNA/DNA is negative
* White blood cell count > 3.5 x 109/L
* Platelets > 150 x 109/L
* Hematocrit > 35%
* Capable of undergoing leukapheresis
* Able to understand and sign informed consent

Donor Exclusion Criteria:

* Psychological traits or psychological or medical conditions which make them unlikely to tolerate the procedure
* Pregnant or lactating female

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lowsky, MD, Principal Investigator — Stanford Medical Center
Locations (1):
- Stanford Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | fTBI/Thiotepa/Fludarabine
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | fTBI/Thiotepa/Fludarabine
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Graft-versus-Host Disease-Free and Relapse-Free Survival (GRFS) Through 1 Year Post-Transplant
Description: The rate of participants who do not experience GvHD and also do not experience relapse are collectively considered to be GRFS. Relapse will be assessed according to the myelodysplastic syndrome or leukemia response criteria. The participants will be assessed for GRFS though 1 year post transplant. The outcome will be reported as the number of participants, a number without dispersion.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | fTBI/Thiotepa/Fludarabine
Number analyzed (Participants) | 7
Participants | 4

2. Secondary Outcome: Number of Participants Experiencing Graft Rejection Through 1 Year Post-Transplant
Description: Graft rejection will be determined on the basis of reaction against the donor hematopoietic cells. The outcome will be reported as the number of participants who experience graft rejection though 1 year post transplant, a number without dispersion
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | fTBI/Thiotepa/Fludarabine
Number analyzed (Participants) | 7
Participants | 0

3. Secondary Outcome: Number of Participants Experiencing Acute Graft-versus-Host Disease (GvHD) Through 1 Year Post-Transplant
Description: The participants will be assessed for acute graft versus host disease (GvHD) though 1 year post transplant. The outcome will be reported as the number of participants who experience acute GvHD, a number without dispersion.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | fTBI/Thiotepa/Fludarabine
Number analyzed (Participants) | 7
Participants | 3

4. Secondary Outcome: Number of Participants With Chronic, Steroid-Requiring Graft-versus-Host Disease (GvHD) Through 1 Year Post-Transplant
Description: The participants will be assessed for chronic, steroid requiring graft versus host disease (GvHD) though 1 year post transplant. The outcome will be reported as the number of participants who experience chronic GvHD, a number without dispersion.
Time Frame: 1 year
Population: The analysis population includes participants who were evaluated for chronic, steroid-requiring GvHD up to 1 year post-transplant. Of the 7 participants initially enrolled, 6 were analyzed for this outcome. One participant was excluded from the analysis due to death from acute GvHD prior to the evaluation of chronic GvHD.
Measure: Number; unit: participants
Arm/Group | fTBI/Thiotepa/Fludarabine
Number analyzed (Participants) | 6
participants | 0

5. Secondary Outcome: Number of Participants With Non-Relapse Mortality Through 1 Year Post-Transplant Without Recurrence of Myelodysplastic Syndrome or Leukemia
Description: Non relapse mortality will be assessed as the number of participants who have died though 1 year post transplant, without a relapse or recurrence of their myelodysplastic syndrome or leukemia. Relapse will be assessed according to the myelodysplastic syndrome or leukemia response criteria. The outcome will be reported as the number of affected participants, a number without dispersion.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | fTBI/Thiotepa/Fludarabine
Number analyzed (Participants) | 7
Participants | 1

6. Secondary Outcome: Number of Participants Who Experience Relapse Through 1 Year Post-Transplant
Description: Relapse will be assessed according to the myelodysplastic syndrome or leukemia response criteria. The outcome will be reported as the number of participants who experience relapse though 1 year post transplant, a number without dispersion.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | fTBI/Thiotepa/Fludarabine
Number analyzed (Participants) | 7
Participants | 0

7. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) will be assessed as the number of participants who remain alive at 1 year post transplant. The outcome will be reported as a number without dispersion.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | fTBI/Thiotepa/Fludarabine
Number analyzed (Participants) | 7
Participants | 6

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | fTBI/Thiotepa/Fludarabine
All-Cause Mortality (participants affected / at risk) | 1/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | fTBI/Thiotepa/Fludarabine (N=7)
Steroid refractory liver GVHD (Hepatobiliary disorders) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | fTBI/Thiotepa/Fludarabine (N=7)
Acute GvHD (Hepatobiliary disorders) | 3 (3)
anal fistula (Gastrointestinal disorders) | 1 (1)
elevated billirubin (Blood and lymphatic system disorders) | 1 (1)
bacteremia (Infections and infestations) | 1 (1)
EBV viremia (Infections and infestations) | 1 (1)
Fungal Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/06/NCT04151706/Prot_SAP_001.pdf